CLINICAL TRIAL: NCT05684679
Title: Efficacy of Incentive Spirometer and Diaphragmatic Breathing Exercise on the Alteration of Arterial Blood Gas Measures in Patients After Coronary Artery Bypass Grafting. A Randomized Comparative Study
Brief Title: Effectiveness of Incentive Spirometer and Diaphragmatic Breathing Exercise on ABG Measures in Post-CABG Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Prinicipal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2019-13
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Post Coronary Artery Bypass Grafting
Keywords: Chest Physiotherapy; Incentive spirometer; Diaphragmatic breathing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IS Group (Experimental): • Patients were instructed to utilize an incentive spirometer in the sitting or half lying position as taught preoperatively.
  * 3 to 5 consecutive breath with the spirometer were interspersed between period of quite breathing.
  * Duration 10-15 minutes/session.
  Interventions: Other: Incentive spirometer plus Chest physiotherapy
- DBE Group (Experimental): • Patients were advised to do diaphragmatic breathing exercise in the sitting or half lying position as taught preoperatively.
  * 3 to 5 consecutive deep breath were interspersed between period of quite breathing.
  * Duration 10-15 minutes/session.
  Interventions: Other: Diaphragmatic breathing exercise plus Chest physiotherapy

INTERVENTIONS:
Other: Incentive spirometer plus Chest physiotherapy — Incentive spirometer was given to IS group. However, a conventional chest physiotherapy was given to both groups in the optimal position.
  Other Names: Huffing, Coughing, Upper and lower limbs active exercises
  Arms: IS Group
Other: Diaphragmatic breathing exercise plus Chest physiotherapy — Diaphragmatic breathing exercise was given to DBE group. In addition, a conventional chest physiotherapy was given in the optimal position.
  Other Names: Huffing, Coughing, Upper and lower limbs active exercises
  Arms: DBE Group

SUMMARY:
The rate of pulmonary complications following Coronary artery bypass graft (CABG) is high. Early pulmonary exercises are important in preventing this complication following cardiac surgery. This study aimed to investigate the effectiveness of incentive spirometer (IS) and diaphragmatic breathing exercise (DBE) on the alteration of arterial blood gas (ABG) measures. The study was based on a two-arm, parallel-group, randomized comparative design. Thirty patients who underwent CABG enrolled in the study based on inclusion and exclusion criteria, randomly allocated into either of the groups, IS Group or DBE Group. IS Group and DBE Group underwent chest physiotherapy with IS and DBE, respectively. ABG measures, including PH of blood, partial pressure of arterial oxygen molecule (PaO2), and partial pressure of arterial carbon dioxide (PaCO2), was assessed using an ABG analyzer at baseline (pre-operation), day1 post-operation, and day2 post-operation. The significance level was kept constant for all statistical analyses at 95%.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) is one of common treatment procedures performed worldwide. Evidence suggest that every year more than 1 million CABG procedure has been performed. Pulmonary complications are one of the most common consequence post CABG.

The incidence of atelectasis after heart operation with cardiopulmonary bypass is still 80-84% in spite of careful fluid & respiratory management. The basic problem in respiratory care of post-surgical patient is atelectasis leading to hypoxemia causing alteration in arterial blood gases (ABGs). Associated with atelectasis are widening alveolar - arterial O2 gradient (as right to left intrapulmonary shunting increases) decrease ventilation perfusion ratio, decrease functional residual capacity and decrease compliance. Chest physiotherapy is routinely used after major abdominal & cardiothoracic surgery to prevent these pulmonary complications following operation.

To date, there is a variable view about the effectiveness of these two primary breathing exercise techniques (incentive spirometer and diaphragmatic breathing exercise). 10-12 Hence an effort to systematically study the effectiveness of these is attempted. Thus, the current study aimed to determine the efficacy of incentive spirometer and diaphragmatic breathing exercises in addition to conventional chest physiotherapy on alteration of ABG measures in patients with post CABG. This study hypothesized that there will be a significant difference between the effect of the IS and DBE on ABG alteration in post CABG patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient with post-CABG,
* Aged between 40 and 60 years,
* Had forced expiratory volume in 1 second (FEV1) <70% of predicted value,
* Showed FEV1/forced vital capacity (FVC) ratio >0.8,
* Weight equal or exceeded the ideal body weight by less than 20%, and
* Patient co-operation.

Exclusion Criteria:

* Aged more than 60 years,
* Weight equal or exceeded the ideal body weight by more than 20%,
* Post-operative respiratory treatment exceeding 20 hours,
* History of Chronic obstructive pulmonary disease (COPD) /thoracic surgery including CABG,
* had thoracic anomalies/unstable angina,
* Developed hemodynamic complication, and
* Non-cooperative/neurological debilitated patient.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-25 (Actual)

PRIMARY OUTCOMES:
PH of Blood | 3 Days
  PH of blood was assessed using an ABG analyzer machine
Partial pressure of Arterial Oxygen molecule (PaO2) | 3 Days
  PaO2 was assessed using an ABG analyzer machine
Partial pressure of Arterial Carbon dioxide molecule (PaCO2) | 3 Days
  PaCO2 was assessed using an ABG analyzer machine

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, MPT, Principal Investigator — King Saud University, Riyadh, Saudi Arabia
Locations (1):
- Rehabilitation Research Chair, Department of Rehabilitation Sciences, king Saud University, Riyadh, Riyadh 11433, Saudi Arabia